CLINICAL TRIAL: NCT02155400
Title: Phase 0 Study of a Thermal Compression Device for Maintenance of Perioperative Normothermia
Brief Title: Thermal Compression Device for Maintenance of Perioperative Normothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Santa Maria, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-28535
Record Dates: First submitted 2014-05-27; First posted 2014-06-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Hypothermia
Keywords: perioperative hypothermia; thermal compression; forced air warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prototype development (Experimental): 10 patients (this phase will be terminated once prototype is confirmed ready) Intervention: prototype device
  Interventions: Device: Prototype / Experimental device
- Treatment arm - Prototype (Active Comparator): - 18 patients Intervention: Prototype device (heating both sole of foot and popliteal fossa with compression)
  Interventions: Device: Prototype / Experimental device
- Control arm - Forced Air Warming Blanket (Active Comparator): 18 patients Intervention: Forced air warming blanket (Bair hugger)
  Interventions: Device: Bair Hugger
- Comparison - Sole of foot only (Active Comparator): 9 patients heating sole of foot only Intervention: prototype device
  Interventions: Device: Prototype / Experimental device
- Comparison - Popliteal fossa only (Active Comparator): 9 patients heating popliteal fossa only Intervention: prototype device
  Interventions: Device: Prototype / Experimental device

INTERVENTIONS:
Device: Bair Hugger — Forced Air Warming Blanket placed over the body of the patient during surgery
  Other Names: Forced Air Warming Blanket
  Arms: Control arm - Forced Air Warming Blanket
Device: Prototype / Experimental device — Contact heating device provides heat to the sole of the foot and popliteal fossa while providing intermittent compression to the lower leg.
  Arms: Comparison - Popliteal fossa only; Comparison - Sole of foot only; Prototype development; Treatment arm - Prototype

SUMMARY:
Getting cold (not maintaining normothermia) around surgery (perioperative period) leads to many negative outcomes for patients including increased wound complications, abnormal heart rhythms and increased blood loss. These all lead to increased length of hospital stay and higher requirements for post operative monitoring. These add to around $3500 of extra costs per patient. The investigators aim to study the effects of a warming device, placed around the patient's legs and/or feet, to determine it's safety, efficacy and eventually compare to the current gold standard of a forced air warming blanket. Forced air warming has been associated with the spread of germs over the surgical field. Hence the need for warming equipment that won't do that.

DETAILED DESCRIPTION:
Cases of inadvertent perioperative hypothermia (IPH) within a hospital setting are often overlooked and should be where the incidence of hypothermia can be eliminated. Heat loss occurs predominantly via convective heat transfer, particularly through glabrous surfaces such as the palms and soles. A decrease in core body temperature can be categorized into mild (32 deg C-36 deg C), moderate (28 deg C-32 deg C), or severe (<28 deg C) hypothermia (2). During preoperative care, patients are dressed solely in a gown and are often exposed to cold waiting areas with little insulation. They are exposed to cold liquids during the wash of the surgical site during sterilization preparation.

Once in the operating room (OR), the patients are naked and exposed to a room temperature well below 36 deg C. To compensate for hypothermia, the hypothalamus attempts to stimulate heat production through sympathetically mediated vasoconstriction, shivering and increased adrenal activity, and through the erection of hair follicles to trap air and retain heat. At the onset of surgery, delivered anesthetics immediately impair the normal autonomic thermoregulatory controls. Colder blood is transferred from the peripheries of the body to the core through a phenomenon known as redistributive hypothermia. Vasodilatation and reduction in muscle tone creates a significant drop in core temperature within the first half-hour of surgery.

IPH is not a rare occurrence. Several sources, including the NICE guidelines, estimate that as many as 70% of patients undergoing normal surgery may be admitted to the Post Anesthesia Care Unit (PACU) hypothermic if the risk is not managed. More conservative estimates put the incidence at 20%. An estimated 48 million inpatient surgical visits were made in the US in 2009, translating to between 10 to 34 million cases of IPH per year in the US alone. All patients are at risk of developing IPH, although certain factors increase the risk of IPH. American Society for Anesthesiology (ASA) grade, lower preoperative temperatures, combined regional and general anesthesia, and intermediate or major surgery are all associated with increased risk of IPH. Under these risk factors, over 17 million patients are at high-risk for becoming hypothermic.

Clinical Impact The development of IPH is strongly correlated with a multitude of physiological organ system changes, impacting the cardiovascular, respiratory, neurologic, immunologic, hematologic, drug metabolic, and wound healing mechanisms. The incidence of several post-surgical complications is increased due to even mild hypothermia (Table 1). Intraoperatively, hypothermia can cause a decrease in cardiac output and heart rate, which can lead to ventricular dysrhythmias. Platelet functions become impaired and there is a decrease in coagulation factors, which lead to greater intraoperative bleeding and blood loss. Hypothermia is associated with a four-fold increase in surgical would infection and twice as many morbid cardiac events.

Overall, compared to non-hypothermic patients, those who suffer IPH experience greater rates of surgical site infections, bleeding, cardiac complications which may require additional monitoring, PACU length of stay, total length of stay, and subjective discomfort. Interestingly, the likelihood of developing hypothermia in an open versus laparoscopic surgery is similar across various types of procedures, most likely attributable to the fact that most laparoscopic procedures are significantly longer when compared to their open surgery counterpart.

Prevention of the effects of redistribution hypothermia is best done before their peripheries become cold, which often occurs before they arrive in the OR. Our audit of Stanford Hospital's Ambulatory Care Centre OR times, from January to March 2013, showed this time was at least 2 hours for all elective patients. Placing responsibility of the device placement on preoperative staff rather than OR staff is also better for compliance, as OR staff are burdened with many other priorities prior to the incision and are more rushed for time.

The critical period to intervene and prevent perioperative hypothermia is in the preoperative phase. This is when peripheral warming can be in place so that when redistribution occurs due to general anesthesia, warm blood flows back from the core rather than cold blood if no peripheral warming is in place. Without preoperative warming, patients will become hypothermic at the beginning of surgery. Intraoperative warming minimizes the extent but does not prevent it.

In one study, 2 cohorts were compared to show the effect on core temperature of preoperative warming to those with no preoperative warming. Both cohorts received intraoperative forced air warming. Without preoperative warming in this cohort, forced air warming methods take 2-5 hours to return the patient to normothermia. Patients cannot leave the PACU hypothermic.

Using a crude works-like prototype the investigators conducted bench testing and collection of preliminary data. In the first hour, no heating was applied followed by two hours with the device turned on. During this time temperature was recorded (oral, arm and leg surface), thermal and general comfort was measured using a visual analogue scale and the presence of shivering or sweating was noted. The device was set up to maintain a maximum at skin temperature of 43°C. This was shown previously to be the higher limit and optimal preoperative warming temperature. This was shown previously to be the higher limit and optimal preoperative warming temperature. The experiment showed that core temperature was maintained in three of the four subjects with one patient becoming hypothermic in the pre device on period. Arm temperature was constant and hypothermic during the experiment. Leg temperature increased with the device on. Thermal comfort and general comfort levels showed the prototype was well tolerated.

The investigators hope to learn from the study:

Prototype development What are the best configurations to apply the device to the patient?

Safety Will the device maintain a consistent temperature at the skin? Will there be no burns occuring? Will the patient not get hyperthermic?

Efficacy Will the device keep the patient from getting cold? If so, what are the relative effects of warming at the soles of the feet and / or with waring at the popliteal fossa? If efficacy is established, is it better than / equivalent to the gold standard of the forced air warming blanket?

Usability Does the device fit into the operative workflow What are the opinions of the users (patients, nurses, doctors) about the usability of the device? Will the device causes patient discomfort while they are awake? Does it improve their thermal comfort?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing procedures with general anesthesia, lasting longer than 30 minutes, that have a leg size that fits a medium sized sequential compression device (DVT leg device) are eligible.

Exclusion Criteria:

* - patients in which procedure hypothermia is desired (eg. some cardiac patients)
* do not have 2 legs for the device to be applied.
* have disease of the legs with altered sensation or may have increased tissue sensitivity to leg warming (peripheral neuropathy, peripheral vascular disease, active legs infections etc)
* patients considered not appropriate by either the attending anesthesiologist or surgeon.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Core temperature | Perioperative period
  average calculated looking for presence of hypothermia (below 36 deg core temp) During surgery, the patient will have their core temperature continuously monitored either via esophageal , tympanic and if available bladder (routine intraoperative monitoring)

SECONDARY OUTCOMES:
Thermal comfort | Measured at 15min intervals in the pre ((within 60 minutes prior to induction of anesthesia) and post op period ((within 60 minutes after awakening from anesthesia)
  measured as visual analogue scale described by patient
General comfort | 15 min intervals in pre ((within 60 minutes prior to induction of anesthesia) and post op period ((within 60 minutes after awakening from anesthesia)
  measured as visual analogue scale, described by patient
Skin injury scale | 15 min intervals during the perioperative period (within 60 minutes prior to induction of anesthesia, during the surgery (expected 3-6 hours) and (within 60 minutes after awakening from anesthesia))
  Presence of skin injury (or impending skin injury) (including burn, abrasion, or tear) scale recorded by research staff.
  -- this would cause the device use to be aborted during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Santa Maria, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hopspital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets

REFERENCES:
- [Derived] Santa Maria PL, Santa Maria C, Eisenried A, Velasquez N, Kannard BT, Ramani A, Kahn DM, Wheeler AJ, Brock-Utne JG. A novel thermal compression device for perioperative warming: a randomized trial for feasibility and efficacy. BMC Anesthesiol. 2017 Aug 11;17(1):102. doi: 10.1186/s12871-017-0395-2. PMID 28800725